CLINICAL TRIAL: NCT02867878
Title: Rapid Recovery of Left Ventricular Function in Patients With Takotsubo Syndrome Undergoing Systemic Infusion of Adenosine: a Randomized Controlled Trial (TITAN Study)
Brief Title: Adenosin to Rapidly Reverse Left Ventricle Impairment in Takotsubo Syndrome
Acronym: TITAN
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: inability to recruiti a sufficient number of patients
Sponsor: University Hospital of Ferrara (Other)
Responsible Party: Principal Investigator, Gianluca Campo, Associate Professor, University Hospital of Ferrara
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 160596
Record Dates: First submitted 2016-08-10; First posted 2016-08-16 (Estimated); Last update posted 2018-10-23 (Actual); Status verified 2018-10

CONDITIONS: Takotsubo Cardiomyopathy; Takotsubo Syndrome
MeSH Terms: conditions — Takotsubo Cardiomyopathy | interventions — Adenosine; Saline Solution

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Adenosine (Experimental): Patients in this arm will receive systemic infusion of adenosine at 140μg/kg/min for 3 minutes plus standard therapy according to current guidelines
  Interventions: Drug: Adenosine
- Saline solution (Placebo Comparator): Patients in this arm will receive systemic infusion of saline solution at 140μg/kg/min for 3 minutes plus standard therapy according to current guidelines
  Interventions: Drug: Saline solution

INTERVENTIONS:
Drug: Adenosine
  Arms: Adenosine
Drug: Saline solution
  Arms: Saline solution

SUMMARY:
The investigators will randomize patients admitted to hospital with Takotsubo diagnosis to systematic high-dose adenosine infusion for 3 minutes (in addition to standard of care) vs. standard of care. The primary aim of the study is to demonstrate that adenosine infusion is associated with a larger and more rapid recovery of left ventricle function.

DETAILED DESCRIPTION:
Takotsubo syndrome is a heart condition that is characterized by the rapid onset of left ventricular dysfunction, usually reversible, and meeting the following diagnostic criteria:

* Transient alterations of regional contractility of the myocardial wall of the right or left ventricle, which are frequently, but not always, preceded by a stressful event (emotional or physical).
* The regional changes in contractility of the myocardial wall, often extend beyond the distribution of a single coronary vessel, and often result in a circumferential ventricular dysfunction of the involved segments.
* Absence of a culprit coronary lesion (eg. Of atherosclerotic plaque rupture, thrombus formation, coronary dissection) or other pathological conditions that may explain the regional changes in contractility of the myocardial wall (eg. Hypertrophic cardiomyopathy, viral myocarditis)
* Reversible electrocardiographic abnormalities of the EKG (ST-T segment elevation or depression, new onset of left bundle branch block, inversion of t wave and / or QTc elongation) during the acute phase (3 months).
* Significant increase in serum natriuretic peptide (BNP or NT-proBNP) during the acute phase
* Troponin significant increase, but relatively small, (disparity between the degree of left ventricular dysfunction and the value of troponin).
* The recovery of left ventricular function during follow-up (3-6 months).

Epidemiology Since the Takotsubo syndrome has been described for the first time in 1991, its incidence, with the passing of years has been increasing, thanks to the possibility with networks for the treatment of acute myocardial infarction, to have a early access to coronary angiography study. Currently this syndrome accounts for 2% of all acute coronary syndromes who are undergoing coronary angiography.

Pathophysiology The pathophysiology of Takotsubo syndrome is complex, and not fully clarified. There are several causes have been suggested over the years to explain the occurrence of this syndrome (vascular and / or myocardial). One of the mechanisms suggested is that there is a systemic response, by the body, to a severe stress which causes a sudden increase of catecholamines endogenous and exogenous; this increase has an effect on the cardiovascular system leading to acute heart failure.

Stress is one of the most common causes behind the onset of this syndrome, and emotional stress (eg. Mourning,quarrel, etc.) and physical (eg. Surgical emergencies, obstetric or psychiatric), but it is not always a present condition.

Recent case reports and clinical studies have shown that patients with this syndrome may experience a reversible damage of the coronary microcirculation, which could be the basis of the important ventricular dysfunction that is observed in these patients. This characteristic may play a significant role in the management of these patients. In fact any targeted therapies to the rapid recovery of the coronary microcirculation function with subsequent improvement in left ventricular function could reduce or prevent the complications related to this case.

Complications During the acute phase of Takotsubo Syndrome the incidence of complications is frequent (18-34% involvement of the right ventricle; obstruction of left ventricular outflow 12-54%; mitral regurgitation 14-25%, 9-20% cardiogenic shock, ventricular thrombus 2-8%, 5-15% atrial fibrillation, ventricular arrhythmias 4-9%, 2-5% bradycardia-asystole) and these complications are often the consequence of left ventricular dysfunction. In fact, the presence of major depression of the ejection fraction (EF) is the main cause of complications in patients with Takotsubo and that the slow pace of recovery of normal EF is closely connected to this risk of complications.

Diagnosis Takotsubo syndrome diagnosis requires, as basic examinations, coronary angiography (allows us to exclude the coronary artery diseases and to highlight the presence of the typical pattern "apical balloon" to the ventriculography) and the echocardiogram ( allow us to highlight the regional alterations of left ventricular kinetics).

Risk Stratification Patients in whom the diagnosis of Takotsubo syndrome is made, they have to be stratified according to their risk profile in patients at high and low risk

Therapy Recently the European Society of Cardiology has prepared a document in which it is suggested therapy to be performed in patients with Takotsubo syndrome according to risk stratification and clinical and echocardiographic data, based on a consensus among the authors in the absence of current randomized clinical studies in support of this strategy.

Mortality The data available report an in-hospital (1-4.5%) and 5 years (3-17%) mortality non-negligible.

Follow-up A recovery of ventricular function is shown at 3-6 months from acute event

Rationale of the study In patients with symptomatic Takotsubo, therapeutic strategies currently used are designed to address, not the pathophysiological mechanism underlying this event, but the complications faced by patients (ie acute heart failure, arrhythmias and hyperkinetic left ventricular thrombosis). No data are currently available about targeted therapies to the treatment of Takotsubo syndrome.

Adenosine is an extracellular signaling molecule that plays a fundamental role in human physiology. Its main effects are: vascular vasodilation, regulation of the activity of the sympathetic nervous system, antithrombotic and regulating blood pressure and heart rate. One of the main uses of adenosine in the cardiovascular field is the production of vasodilation of the coronary microcirculation to produce hyperemia, as for example in the assessment of intermediate coronary stenoses using fractional flow reserve (FFR). It also finds use even in the course of acute myocardial infarction in reducing the phenomenon of slow-flow in the course of primary angioplasty, even if the results of the studies currently available are not unambiguous interpretation.

Galiuto et al. have demonstrated that, regardless of the underlying etiology, in patients with Takotsubo syndrome, it shows the presence of an acute and reversible vasoconstriction of the coronary microcirculation, which may represent a common pathophysiologic mechanism in these patients. In the study the investigators underline also as the use of a systemic infusion of adenosine at a dose of 140 micrograms / kg / min for 90 seconds determines an initial improvement, statistically significant, of the left ventricular function in these patients. The study was observational, and have not been taken into consideration clinical outcomes.

Numerous studies performed in patients with STEMI (ST-segment elevation myocardial infarction) have shown that the adenosine infusion systems, although at high doses, causes only mild adverse effects (es. dyspnea, chest pain, transient ventricular atrium block, hypotension ) and all quick resolution with the suspension of the infusion.

Objective of the study The objective of this study is to demonstrate that in patients with Takotsubo syndrome diagnosis, the use of adenosine infusion at high doses, immediately after the diagnosis of disease, and the absence of documentation of coronary artery disease, it is able to enhance the EF of these patients to 48 hours after diagnosis, compared with standard therapy.

Study Design It is an multicenter, randomized, single-blind study, phase IIa.

Once coronary angiography demonstrated the absence of coronary artery disease and confirmed the diagnosis of Takotsubo syndrome patients will undergo a baseline echocardiography and then randomized, using a randomization system electronic, 1: 1 to receive:

* Systemic infusion of adenosine to 140μg / kg / min for 3 minutes + standard therapy
* Placebo (saline to 3 minutes) + standard therapy

Randomization will be stratified by the following variables:

* gender (male vs. female)
* age (<65 years vs. ≥65 years) The standard therapy, will be allocated based on the risk stratification of patients enrolled. Patients will then be assessed by echocardiography at 24 hours, 48 hours and 1 month according to the parameters given in the echocardiographic analysis section.

All patients will be followed up with clinical follow-up up to one year.

PRESPECIFIED SUBSTUDY As has been shown in previous studies, patients with Takotsubo syndrome have reversible coronary microvascular damage.

The purpose of our study is to assess whether the infusion of high-dose adenosine e.v favors the improvement of left ventricular ejection function quickly.

With this sub-study we want to evaluate, also, if there is also in our series a damage of the coronary microcirculation.

Patients participating in the sub-study, randomized in the Adenosine arm, the evaluation of coronary microcirculation will be performed by calculating the IMR (microcirculatory resistance index) during the infusion of adenosine required by randomization.

The IMR is a validated method for measuring the function of the coronary microcirculation. By using a previously positioned guide pressure on the left anterior descendent (LAD) coronary artery, IMR is evaluated by the thermodilution technique analyzing the transit time of a predetermined quantity (3 ml) of saline at room temperature injected into the coronary artery.

3 consecutive injection of 3 mL of saline solution are performed at baseline, and evaluated the average transit time for resting (Tmn). Later, during maximal hyperemia induced by systemic infusion of Adenosine a140μg / kg / min, 3 new injections of saline at room temperature are performed, and the mean transit temple during hyperemia (Tmnhyp) is measured. Tmnhyp multiplying by the average value of distal coronary pressure (Pd) registered during maximal hyperemia, get the IMR value (IMR: Tmnhyp x Pd) which is considered in the normal range if less than 25. A value above 25 indicates the presence of a damage of the coronary microcirculation.

ELIGIBILITY:
Inclusion Criteria:

* 18 years old
* Evidence of typical anatomical pattern to the left ventriculography (total akinesia of the mid-apical segments with hypercontractility basal segments) associated with the presence of criteria for the diagnosis of Takotsubo syndrome (Table 1)
* signing of informed consent

Exclusion Criteria:

* allergy to adenosine
* known and documented diagnosis of asthma
* pre-existing ischemic heart disease
* presence of arrhythmic complication (AV block grade II type 2 and third degree)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2016-08 (Actual); Primary Completion 2018-10 (Actual); Study Completion 2018-10 (Actual)

PRIMARY OUTCOMES:
left ventricle ejection fraction (%) | 48 hours
  an indipendent corelab will review all images from 48-hour ecocardiography to establish LVEF value (%)

SECONDARY OUTCOMES:
left ventricle ejection fraction (%) | 24 hours
  an indipendent corelab will review all images from 24-hour ecocardiography to establish LVEF value (%)
left ventricle ejection fraction (%) | 1 month
  an indipendent corelab will review all images from 1-month ecocardiography to establish LVEF value (%)
wall motion score index | 24 hours
  an indipendent corelab will review all images from 24-hour ecocardiography to calculate WMSI value (number)
wall motion score index | 48 hours
  an indipendent corelab will review all images from 48-hour ecocardiography to calculate WMSI value (number)
wall motion score index | 1 month
  an indipendent corelab will review all images from 1-month ecocardiography to calculate WMSI value (number)
acute heart failure | 1 month
  it is defined as dyspnea + crackles on auscultation + signs on X-ray of chest congestion
intravenous diuretics | 1 month
  it is defined as the total count of mg of furosemide
emergency room admission | 1 month
  Access to the emergency room for dyspnea/heart failure
major adverse events | 1 year
  cumulative incidence of all-cause death and hospital admission for cardiovascular causes
hypokinetic arrhythmias | 1 hour
  cumulative occurrence of hypokinetic arrhythmias (asystole, atrio-venticular block) in the course of administration of adenosine as shown by electrocardiogram recording
arterial hypotension | 1 hour
  persistent hypotension (arterial blood pressure <90 mmHg) during administration of adenosine as shown by invasive blood pressure recording
side effects | 1 hour
  Persistent symptoms (nausea, dyspnea, hot flush, etc.) that require premature discontinuation of the administration of adenosine

CONTACTS AND LOCATIONS:
Overall Officials: Matteo Tebaldi, MD, Principal Investigator — Azienda Ospedaliera Universitria di Ferrara
Locations (1):
- University Hospital of Ferrara, Cona, Ferrara, Italy

IPD SHARING:
Plan to Share IPD: Undecided